CLINICAL TRIAL: NCT00558779
Title: Surgical Manipulation of the Ascending Aorta and Cerebral Infarction Following CABG
Brief Title: Surgical Manipulation of the Aorta and Cerebral Infarction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49/07; F/13/03
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Heart Disease; Stroke; Cerebral Infarction
Keywords: Coronary artery bypass; off pump coronary artery bypass grafting (OPCAB)
MeSH Terms: conditions — Coronary Disease; Stroke; Cerebral Infarction | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: OBCAB (Off Pump Coronary Artery Bypass Grafting)
- 2 (Active Comparator)
  Interventions: Procedure: CABG (coronary artery bypass grafting)

INTERVENTIONS:
Procedure: OBCAB (Off Pump Coronary Artery Bypass Grafting) — OPCAB with sparing of aortic manipulation (eg, no aortic cannulation for cardiopulmonary bypass, no aortic cross-clamp, no side-clamping of the aorta). Graft anastomosis to the central circulation with y-grafts on the arteria thoracica interna or on the aorta with help of the Heart-string-system (Guidant)
  Arms: 1
Procedure: CABG (coronary artery bypass grafting) — conventional CABG with cardiopulmonary bypass
  Arms: 2

SUMMARY:
The purpose of the study is to compare two surgical strategies for coronary artery bypass grafting with respect to the occurrence of cerebral infarctions made visible by magnetic resonance imaging

DETAILED DESCRIPTION:
Stroke is one of the most devastating complications following coronary artery bypass grafting (CABG) with an overall incidence ranging from 2.0 % to 3.2 %. The presumed etiology for the majority of strokes after CABG is atheroembolism from the diseased aorta ascendens caused by surgical manipulation. Off-pump coronary artery bypass grafting (OPCAB) allows the construction of bypass grafts without surgical manipulation of the aorta. Yet a trial comparing different surgical strategies with stroke as the primary end point would require several thousand patients to achieve an adequate statistical power. The number of patients can be substantially reduced, if cerebral damage is assessed by diffusion-weighted magnetic resonance imaging (DW-MRI). Using DW-MRI we have recently demonstrated that 25% of a patient population undergoing CABG without an increased risk of stroke showed new cerebral infarctions. These new cerebral lesions all showed an embolic pattern, became visible at T2-weighted images and were clinically silent, e .g. did not cause a new focal neurologic deficit. Given the much higher frequency of cerebral lesions assessed by DW-MRI than clinically apparent stroke, DW-MRI is an ideal surrogate parameter for the assessment of cerebral damage in patients undergoing CABG.

The aim of the study is therefore, to investigate the influence of the surgical technique on the occurence of new ischemic cerebral lesions as assessed by DW-MRI in patients undergoing CABG in a prospective randomized setting. We hypothesize that OPCAB, which enables sparing of aortic manipulation, will reduce cerebral infarctions in patients with an increased risk for perioperative stroke.

ELIGIBILITY:
Inclusion Criteria:

* age > 72
* history of stroke
* cerebrovascular artery disease with stenosis > 50%
* peripheral arterial disease.

Exclusion Criteria:

* urgent or emergency operation
* unstable angina
* reoperation
* concomitant valvular disease requiring surgery
* implanted pacemaker or other incorporated ferromagnetic material
* claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-11; Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
occurrence and number of cerebral infarctions assessed by magnetic resonance imaging | 2-7 days after surgery

SECONDARY OUTCOMES:
mortality | within hospital stay following surgery
stroke | within hospital stay following surgery
delirium | within hospital stay following surgery
neurocognitive performance | within hospital stay following surgery
multi-organ failure | within hospital stay following surgery
myocardial infarction | within hospital stay following surgery
completeness of revascularisation | within hospital stay following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wilko Reents, MD, Principal Investigator — Department of Cardiothoracic Surgery
Locations (1):
- Department of Cardiothoracic Surgery, University Hospital Wuerzburg, Würzburg, Germany

REFERENCES:
- [Background] Stamou SC, Hill PC, Dangas G, Pfister AJ, Boyce SW, Dullum MK, Bafi AS, Corso PJ. Stroke after coronary artery bypass: incidence, predictors, and clinical outcome. Stroke. 2001 Jul;32(7):1508-13. doi: 10.1161/01.str.32.7.1508. PMID 11441193
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Calafiore AM, Di Mauro M, Teodori G, Di Giammarco G, Cirmeni S, Contini M, Iaco AL, Pano M. Impact of aortic manipulation on incidence of cerebrovascular accidents after surgical myocardial revascularization. Ann Thorac Surg. 2002 May;73(5):1387-93. doi: 10.1016/s0003-4975(02)03470-7. PMID 12022522
- [Background] Sellke FW, DiMaio JM, Caplan LR, Ferguson TB, Gardner TJ, Hiratzka LF, Isselbacher EM, Lytle BW, Mack MJ, Murkin JM, Robbins RC; American Heart Association. Comparing on-pump and off-pump coronary artery bypass grafting: numerous studies but few conclusions: a scientific statement from the American Heart Association council on cardiovascular surgery and anesthesia in collaboration with the interdisciplinary working group on quality of care and outcomes research. Circulation. 2005 May 31;111(21):2858-64. doi: 10.1161/CIRCULATIONAHA.105.165030. PMID 15927994
- [Background] Bendszus M, Reents W, Franke D, Mullges W, Babin-Ebell J, Koltzenburg M, Warmuth-Metz M, Solymosi L. Brain damage after coronary artery bypass grafting. Arch Neurol. 2002 Jul;59(7):1090-5. doi: 10.1001/archneur.59.7.1090. PMID 12117356